CLINICAL TRIAL: NCT02481206
Title: Wearable Cardioverter Defibrillator in Hemodialysis Patients (WED-HED) Study
Acronym: WED-HED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subject enrollment
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90D0126
Record Dates: First submitted 2015-06-08; First posted 2015-06-25 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Sudden Cardiac Death; Sudden Cardiac Arrest
Keywords: Ventricular Tachycardia
MeSH Terms: conditions — Death, Sudden, Cardiac; Tachycardia, Ventricular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wearable Cardioverter Defibrillator (Experimental): End Stage Renal Disease (ESRD) patients beginning hemodialysis will use a Wearable Cardioverter Defibrillator for six months
  Interventions: Device: Wearable Cardioverter Defibrillator
- Conventional Treatment (No Intervention): Conventional Treatment

INTERVENTIONS:
Device: Wearable Cardioverter Defibrillator — Wearable Cardioverter Defibrillator
  Other Names: WCD; LifeVest
  Arms: Wearable Cardioverter Defibrillator

SUMMARY:
A multi-center, prospective, randomized controlled clinical trial with 1:1 assignment of treatment and control. This study will evaluate the impact of wearable cardioverter defibrillator use on sudden cardiac death in incident hemodialysis patients. The study will enroll up to 2,600 subjects. A maximum of 200 sites in the USA will be used for enrollment.

DETAILED DESCRIPTION:
Objective:

To study the impact of wearable cardioverter defibrillator (WCD) use on sudden cardiac death in hemodialysis patients.

Study Population:

Participants will be patients beginning hemodialysis (<2 months from initiation) who are ≥ 50 years old.

Intervention:

A WCD will be used for protection against sudden cardiac death (SCD).

Study Design:

The study will be a multi-center, prospective, randomized controlled trial with 1:1 assignment of treatment and control.

Study Size:

The study will enroll up to 2,600 subjects. A maximum of 200 sites will be used for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease (ESRD) requiring hemodialysis
* On hemodialysis for ≤ 2 calendar months or scheduled to begin hemodialysis within 1 calendar month
* ≥50 years of age
* Documented Ejection Fraction > 35% within the previous calendar year
* - If the patient has been hospitalized for a myocardial infarction or heart failure decompensation, the Ejection Fraction measurement must have occurred during the last hospitalization or after discharge

Exclusion Criteria:

* Is receiving or will receive hemodialysis due to acute kidney injury and is not expected to receive subsequent chronic hemodialysis therapy
* Patient has an active ICD
* Patient has a unipolar pacemaker
* Patient has physical or mental conditions preventing him/her from interacting with or wearing a Wearable Cardioverter Defibrillator
* Patient has a chest circumference at the level of the xiphoid of < 24 inches
* Patient has a chest circumference at the level of the xiphoid of > 56 inches
* Patient has an advance directive prohibiting resuscitation
* Patient has cancer or other terminal disease (excluding ESRD) with expected survival less than 6 months
* Patient is medically unstable for reasons not specifically related to kidney disease
* Patient is scheduled for live-donor kidney transplantation within 6 calendar months
* Patient is unable to consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Zareba, M.D., Ph.D, Principal Investigator — University of Rochester; Charles A. Herzog, M.D., Principal Investigator — Chronic Disease Research Group, Hennepin County Medical Center, University of Minnesota
Locations (31):
- United States (31):
  - Corona, California
  - Downey, California
  - Escondido, California
  - Los Angeles, California
  - Sacramento, California
  - San Dimas, California
  - San Luis Obispo, California
  - Whittier, California
  - Stamford, Connecticut
  - Hialeah, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Winter Garden, Florida
  - Albany, Georgia
  - Columbus, Georgia
  - Fort Wayne, Indiana
  - Greenbelt, Maryland
  - Detroit, Michigan
  - Rochester Hills, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - The Bronx, New York
  - Durham, North Carolina
  - Canton, Ohio
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Houston, Texas
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study began on 30-Jun-2015 and ended 15-Feb-2017. Subjects beginning or anticipated to begin dialysis were recruited from kidney clinics and dialysis centers.
Pre-assignment Details: Since the sudden death rate is highest early after initiating hemodialysis, subjects could be enrolled from 1 month before starting dialysis to 2 months after. All subjects had to have a left ventricular ejection fraction over 50%. Subjects were shown a wearable defibrillator and were anticipated to be able to use it prior to enrollment.
Groups:
- Wearable Cardioverter Defibrillator: End Stage Renal Disease (ESRD) patients beginning hemodialysis will use a Wearable Cardioverter Defibrillator for six months, in addition to conventional treatment.
- Conventional Treatment: End Stage Renal Disease (ESRD) patients beginning hemodialysis will get conventional treatment only.
Period: Overall Study
Arm/Group | Wearable Cardioverter Defibrillator | Conventional Treatment
Started | 34 | 32
Completed | 29 | 31
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Conventional Treatment: Conventional treatment during hemodialysis initiation will be applied to this arm.
- Total: Total of all reporting groups
Arm/Group | Wearable Cardioverter Defibrillator | Conventional Treatment | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.6) | 60.1 (9.5) | 59.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data entry error on one subject in control group.
  Participants
    number analyzed (Participants) | 34 | 31 | 65
    Female | 14 | 9 | 23
    Male | 20 | 22 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hypertension [Count of Participants; unit: Participants] | 34 | 32 | 66
Diabetes [Count of Participants; unit: Participants] | 28 | 24 | 52
History of Heart Failure [Count of Participants; unit: Participants] — Population: Missing data on 3 WCD subjects and 1 Control subject
  Participants
    number analyzed (Participants) | 31 | 31 | 62
    (all) | 9 | 9 | 18
Previous Myocardial Infarction [Count of Participants; unit: Participants] — Population: Missing data on 2 WCD subjects and 3 Control subjects
  Participants
    number analyzed (Participants) | 32 | 29 | 61
    (all) | 5 | 1 | 6
History of Ventricular Arrhythmias [Count of Participants; unit: Participants] — Population: Missing data on 2 Control subjects
  Participants
    number analyzed (Participants) | 34 | 30 | 64
    (all) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Sudden Cardiac Death (SCD) Mortality as Assessed by Intention-to-Treat Analysis
Description: This is an intention to treat analysis of SCD, with subjects analyzed by randomization assignment regardless of treatment crossovers or noncompliance. For witnessed deaths, SCD will be defined as an unexpected, non-traumatic, non-self-inflicted fatality in otherwise stable subjects who die within one hour of the onset of the terminal symptoms (dialysis noncompliance or withdrawal subjects excluded). Subjects dying more than one hour after a sudden cardiac arrest from a ventricular arrhythmia will be designated as non-sudden death due to ventricular arrhythmia. For unwitnessed deaths, if the subject is found dead within 24 hours of being well the death will be designated as SCD. If more than 24 hours has passed the death will be designated as indeterminate.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Wearable Cardioverter Defibrillator | Conventional Treatment
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

2. Secondary Outcome: Total Mortality
Description: All cause mortality
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Wearable Cardioverter Defibrillator | Conventional Treatment
Number analyzed (Participants) | 29 | 31
Participants | 0 | 0

3. Secondary Outcome: Sudden Cardiac Death (SCD) Mortality Assessed by As-treated Analysis
Description: This is an as-treated analysis of SCD. For witnessed deaths, SCD will be defined as an unexpected, non-traumatic, non-self-inflicted fatality in otherwise stable subjects who die within one hour of the onset of the terminal symptoms (dialysis noncompliance or withdrawal subjects excluded). Subjects dying more than one hour after a sudden cardiac arrest from a ventricular arrhythmia will be designated as non-sudden death due to ventricular arrhythmia. For unwitnessed deaths, if the subject is found dead within 24 hours of being well the death will be designated as SCD. If more than 24 hours has passed the death will be designated as indeterminate.
Time Frame: 6 months
Population: To allow for crossovers, the analysis unit is patient months. Note: There were crossover months in the treatment group that were included in the control group for this as-treated analysis. That is, since all WCD users had months during which they did not use a WCD, they are also counted in the WCD not used group.
Measure: Mean (95% Confidence Interval); unit: patient months
Units Other Than Participants: patient months
Groups:
- Wearable Cardioverter Defibrillator Used: Time during which a wearable defibrillator was actually worn, whether in the intention to treat wearable defibrillator arm or the control arm (crossovers). All other time will be analyzed as part of the control group.
- Wearable Cardioverter Defibrillator Not Used: Time during which a wearable defibrillator was not worn, whether in the intention to treat wearable defibrillator arm (crossovers) or the control arm.
Arm/Group | Wearable Cardioverter Defibrillator Used | Wearable Cardioverter Defibrillator Not Used
Number analyzed (Participants) | 29 | 60
Number analyzed (patient months) | 40 | 320
patient months | 0 [0 to 0.088] | 0 [0 to 0.012]

4. Secondary Outcome: Clinical Status of Sudden Cardiac Arrest (SCA) Survivors
Description: This is an intention to treat analysis of the clinical status of participants who experience an SCA and survive at least 48 hours, as determined by the Glasgow Coma Scale (numeric scale is 3 to 14, higher is better).
Time Frame: 48 hours after SCA
Population: Study participants from both arms who experienced SCA.
Arm/Group | Wearable Cardioverter Defibrillator | Conventional Treatment
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Potentially Life Threatening Arrhythmias
Description: In the Wearable Cardioverter Defibrillator arm, determine the incidence of potentially life-threatening arrhythmias while the device was worn. Life-threatening arrhythmias are defined as ventricular tachycardia over 150 beats per minute and ventricular fibrillation (VTVF).
Time Frame: 6 months
Population: All subjects using a wearable cardioverter defibrillator were included (treatment group assignment and crossovers from control group assignment). Only months with wearable cardioverter defibrillator use were used for calculations.
Measure: Mean (90% Confidence Interval); unit: VTVF per patient-month
Units Other Than Participants: patient-months
Arm/Group | Wearable Cardioverter Defibrillator
Number analyzed (Participants) | 29
Number analyzed (patient-months) | 40
VTVF per patient-month | 0 [0 to 0.098]

6. Secondary Outcome: Risk of Inappropriate Therapy
Description: Device reported inappropriate shocks/treatments during patient wear time in experimental device wearing arm
Time Frame: 6 months
Population: as for outcome 5
Measure: Mean (90% Confidence Interval); unit: inappropriate shocks per patient month
Units Other Than Participants: patient months
Arm/Group | Wearable Cardioverter Defibrillator
Number analyzed (Participants) | 29
Number analyzed (patient months) | 40
inappropriate shocks per patient month | 0 [0 to 0.098]

7. Secondary Outcome: Compliance With Wearable Cardioverter Defibrillator Therapy
Description: In the group randomized to receive a Wearable Cardioverter Defibrillator, the device recorded time of use will be used to determine compliance measured as a % of time available for use.
Time Frame: 6 months
Population: All trial participants who were randomized to wear a wearable cardioverter defibrillator.
Measure: Mean (Standard Deviation); unit: Percentage of time available for use
Arm/Group | Wearable Cardioverter Defibrillator
Number analyzed (Participants) | 29
Percentage of time available for use | .23 (.33)

8. Secondary Outcome: Kidney Disease Quality of Life 36-item Short Form Survey (KDQOL-36) As Assessed by As-treated Analysis at 2 Months
Description: A self completed questionnaire, the KDQOL-36 has five scales scored from 0 to 100, with higher numbers considered better (i.e., better health related quality of life). For reporting the total score, the 5 scales were averaged for each subject, creating a 0 to 100 range with higher scores considered better.
Time Frame: 2 months
Population: All subjects completing the KDQOL-36 at 2 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wearable Cardioverter Defibrillator | Conventional Treatment
Number analyzed (Participants) | 25 | 28
units on a scale | 79.6 (10.6) | 82.7 (9.1)

9. Secondary Outcome: Kidney Disease Quality of Life 36-item Short Form Survey (KDQOL-36) As Assessed by As-treated Analysis at 6 Months
Description: as for outcome 8
Time Frame: 6 months
Population: All subjects completing the KDQOL-36 at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wearable Cardioverter Defibrillator | Conventional Treatment
Number analyzed (Participants) | 16 | 15
units on a scale | 79.9 (12.4) | 83.4 (11.7)

ADVERSE EVENTS:
Time Frame: 6 months
Description: An unanticipated adverse device effect is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.
Arm/Group | Wearable Cardioverter Defibrillator | Conventional Treatment
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 5/29 | 0/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wearable Cardioverter Defibrillator (N=29) | Conventional Treatment (N=31)
Discomfort (Skin and subcutaneous tissue disorders) | 4 | 0 (0) — Discomfort with wearing the device
Frequent false alarms (Social circumstances) | 1 | NA — study withdrawal due to self-terminating arrhythmia alarms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT02481206/Prot_SAP_000.pdf